CLINICAL TRIAL: NCT06596291
Title: First-In-Human Phase 1b/2a Dose Escalation Study of EG110A, Administered by Intradetrusor Injections to Adult Participants With Neurogenic Detrusor Overactivity-related Incontinence Following Spinal Cord Injury Who Regularly Perform Clean Intermittent Catheterization
Brief Title: Dose Escalation Study of EG110A, Administered by Intradetrusor Injections to Adults With Neurogenic Detrusor Overactivity-related Incontinence Following Spinal Cord Injury Who Regularly Perform Clean Intermittent Catheterization
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EG 427 (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EG110A-001-01; HT94252510505_CDMRP (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Neurogenic Detrusor Overactivity; Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This first-in-human clinical study, performed in SCI participants with UI due to NDO and an inadequate response to current therapy, will evaluate the safety and tolerability of EG110A, and explore the potential doses for further clinical development. The present clinical study will also investigate the efficacy of EG110A via data collected in a bladder diary and via urodynamic assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EG110A (low dose) (Experimental): Patients who Received EG110A (low dose)
  Interventions: Drug: EG110A
- EG110A (Middle Dose) (Experimental): Patients who Received EG110A (middle dose)
  Interventions: Drug: EG110A
- EG110A (High Dose) (Experimental): Patients who Received EG110A (high dose)
  Interventions: Drug: EG110A

INTERVENTIONS:
Drug: EG110A — Participants treated with EG110A

SUMMARY:
This is a first-in-human, Phase 1b/2a, open-label, dose-escalation study of a single treatment course consisting of multiple intradetrusor injections of EG110A in male and female adult participants with Neurogenic Detrusor Overactivity (NDO)-related incontinence following Spinal Cord Injury (SCI), who have persistent incontinence after standard of care therapy and who perform Clear Intermittent Catheterization (CIC) on a regular basis.

DETAILED DESCRIPTION:
This first-in-human clinical study, performed in SCI participants with Urinary Incontinence (UI) due to NDO and an inadequate response to current therapy, will evaluate the safety and tolerability of EG110A, and explore the potential doses for further clinical development. The present clinical study will also investigate the efficacy of EG110A via data collected in a bladder diary and via urodynamic assessments.

ELIGIBILITY:
Main Inclusion Criteria:

1. Participant has stable supra-sacral traumatic SCI with American Spinal Injury Association (ASIA) Impairment Scale grade A, B, C, D or E which occurred at least 12 months before Screening.
2. Participant has UI due to urodynamically-confirmed NDO for at least 3 months prior to Screening.
3. Participant has:

   1. been treated for NDO for at least 3 months prior to Screening with an adequate course of oral pharmacotherapy(ies) and/or has had intolerable side-effects and/or exhibited an inadequate response in the opinion of the investigator and participant, i.e., at least 8 UI episodes in a week despite consistent use of the therapy. Participant does not wish to proceed to BoNT/A treatment, and their next step would be surgical intervention.

      OR
   2. had an inadequate response to BoNT/A treatment in the opinion of the investigator and participant, i.e., at least 8 UI episodes in a week, and the last BoNT/A treatment for their NDO was at least 6 months prior to screening. Treatment with BoNT/A was not started more than 7 years ago, and their next step would be surgical intervention.

Main Exclusion Criteria:

1. Participant has previous or current tumor or malignancy affecting the spinal column or spinal cord, or any other nonstable cause of SCI.
2. Participant with active oral or genital herpes lesion. If the participant has an active oral or genital herpes infection this needs to be treated and healed first. The participant may be rescreened once the lesion has fully healed (at least 4 weeks after the lesion has healed).
3. Participant had cancer therapy or radiotherapy ≤ 4 weeks prior to Screening and has toxicities/AEs attributable to previously administered cancer therapies that have not resolved or stabilized.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | 1 year
  Any participant who has a reported treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Urodynamic variables: changes at Weeks 12 and 52 compared to baseline | 1 year
  Changes in urodynamic variables will be assessed at Weeks 12 and 52.
Bladder Diary measures: changes in 7 days' mean daily episodes at Weeks 12 and 52 compared to baseline | 1 year
  7 day bladder diary with recording of urinary incontinence episodes, daily catheterization rates, and volume per catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Haag-Molkenteller, MD, Study Director — EG 427
Locations (4):
- United States (4):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Sidney Kimmel Medical College, Philadelphia, Pennsylvania
  - UTHealth Houston / TIRR Memorial Hermann, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more about the clinical study EG110A-001-01 — https://clinicaltrials.eg427.com/